CLINICAL TRIAL: NCT00497874
Title: An Expert System to Reduce Depression in Primary Care
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pro-Change Behavior Systems (Other)
Collaborators: Harvard Vanguard Medical Associates (Other); Cook County Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R44MH060522 (NIH)
Record Dates: First submitted 2007-07-05; First posted 2007-07-09 (Estimated); Results first posted 2015-07-07 (Estimated); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Depression; Depressive Disorder, Major
Keywords: depression; stage of change; intervention; randomized clinical trial; population-based; expert system
MeSH Terms: conditions — Depression; Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Computer-tailored intervention (Experimental): Stage-based manual and three computer-tailored reports
  Interventions: Behavioral: Computer-tailored intervention
- Usual care (No Intervention): Usual primary care treatment

INTERVENTIONS:
Behavioral: Computer-tailored intervention — Stage-based manual and three computer-tailored reports
  Other Names: Roadways to Healthy Living
  Arms: Computer-tailored intervention

SUMMARY:
The purpose of this study is to determine whether a home-based intervention matched to stage of change (readiness) for using effective methods to prevent or reduce depression can improve depression outcomes in primary care.

DETAILED DESCRIPTION:
A variety of effective interventions exist for people who are willing to seek help for depression. However, there is a lack of interventions for individuals who are not willing to seek help or follow through with treatment recommendations. This is the first population-based intervention for depression that is appropriate for individuals in all stages of change-not merely the minority who are prepared to take action. Two primary care samples were included: 1) patients at risk for or experiencing depression but not involved in or planning treatment (Untreated Sample), and 2) patients newly prescribed antidepressant medication (Antidepressant Sample). Patients from both samples were randomly assigned to receive the intervention consisting of telephone assessments, a stage-based workbook, and three individualized, computer-generated reports mailed to the home (n=443), or usual care (n=459). Primary outcomes, assessed at 9 months, were change in depression severity, reliable and clinically significant change in depression severity, stage of change for using effective methods or prevent or reduce depression, onset of major depression if experiencing only subclinical symptoms at baseline, and medication adherence. The study design included an examination of whether the intervention effect was moderated by primary care sample, baseline use of effective methods to prevent or reduce depression, and level of depression.

ELIGIBILITY:
Inclusion Criteria:

* At risk for or experiencing depression (i.e., Beck Depression Inventory-II (BDI) score of 10 or higher; current major depression, minor depression, or dysthymia; or past major depression, minor depression, or dysthymia)

Exclusion Criteria:

* Younger than age 18
* Involved in counseling or planning counseling in the next 30 days
* Taking antidepressant medication or planning to take antidepressants in the next 30 days (exclusion criterion for Untreated Sample only)
* Suicidal ideation
* Severe depression (BDI > 28) and deemed inappropriate for study by site clinician
* BDI <10 and in the Maintenance stage for using effective methods to prevent or reduce depression
* History of bipolar disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 902 (Actual)
Dates: Start 2003-07; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah A. Levesque, Ph.D., Principal Investigator — Pro-Change Behavior Systems, Inc.
Locations (2):
- United States (2):
  - John H. Stroger Hospital, Chicago, Illinois
  - Harvard Vanguard Medical Associates, Newton, Massachusetts

REFERENCES:
- [Result] Levesque DA, Van Marter DF, Schneider RJ, Bauer MR, Goldberg DN, Prochaska JO, Prochaska JM. Randomized trial of a computer-tailored intervention for patients with depression. Am J Health Promot. 2011 Nov-Dec;26(2):77-89. doi: 10.4278/ajhp.090123-QUAN-27. PMID 22040388

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 902 primary care patients were recruited from the 17 clinics of a large multi-specialty medical group practice in Eastern Massachusetts (N=791) and a large health center in Chicago (N=111).
Groups:
- Intervention: Stage-based manual and three computer-tailored reports
Period: Overall Study
Arm/Group | Intervention | Usual Care
Started | 443 | 459
Completed | 296 | 343
Not Completed | 147 | 116
Not completed — Withdrawal by Subject | 48 | 17
Not completed — Illness | 8 | 4
Not completed — Death | 2 | 4
Not completed — Unable to contact | 52 | 67
Not completed — Unable to schedule | 37 | 24

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Usual Care | Total
Number analyzed (Participants) | 443 | 459 | 902
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 391 | 408 | 799
  >=65 years | 52 | 51 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.0 (14.7) | 47.1 (15.3) | 47.5 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 308 | 314 | 622
  Male | 135 | 145 | 280
Region of Enrollment [Number; unit: participants]
  United States | 443 | 459 | 902

OUTCOME MEASURES:

1. Primary Outcome: Change in Depression Severity
Description: Depression was assessed using the Beck Depression Inventory, 2nd Edition (BDI-II)(Beck, Steer, & Brown, 1996). In this self-report measure, 21 symptoms of depression are rated on a 0-3 scale. Scores for the 21 items are summed to yield a total score ranging from 0 to 63. The change scores reported here are the difference between the total BDI-II scores at baseline and 9 months (i.e., 9 months minus baseline). Change scores range from -63 to +63, with larger negative scores indicating greater reduction in depression.
Time Frame: Baseline, 9 months
Population: Multiple imputation
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Intervention: Usual primary care + computer-tailored intervention
- Usual Care: Usual primary care
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 443 | 459
units on a scale | -5.4 (8.8) | -3.7 (7.5)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Multiple imputation was used to estimate missing data for the 9-month assessment. Ten datasets were imputed using Multivariate Imputation by Chained Equations. Using SAS v9.1 PROC MI, the complete datasets were analyzed using complete data methodology-in this case, the t-test-and the results pooled; Test type: Non-Inferiority or Equivalence — Power analysis shows that sample size provided power of at least .80 to detect estimated differences; p = .003, t-test, 1 sided — Statistical significance of the pooled results was evaluated using a t-test and degrees of freedom that take into account the uncertainty in the data and the uncertainty due to missing values; t(145) = 2.8

2. Secondary Outcome: Number of Participants Exhibiting a Reliable and Clinically Significant Change in Depression Severity
Description: Two statistical criteria (Jacobson & Truax, 1991a; Atkins, Bedics, McGlinchey, & Beauchaine, 2005) were used to define reliable and clinically significant improvement. The first involved selecting a cutoff that represents remission or the absence of symptoms, which was selected to be BDI-II < 9. The second involved selecting a pre-post difference score that represents a statistically reliable change (e.g., how much change-1 point, 5 points, 10 points-is needed to be 95% confident that a real change has occurred, rather than just a chance fluctuation due to the unreliability of the measure?) Using a general formula for calculating reliable change that incorporates test-retest reliability (Jacobson & Truax, 1991b), reliable change for the BDI-II was calculated to be 5.13, and rounded down to 5. Thus, reliable and clinically significant improvement on the BDI-II was defined as a reduction of 5 or more points from baseline to follow-up and a follow-up score < 9.
Time Frame: 9 months
Population: Multiple imputation
Measure: Number; unit: Participants
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 443 | 459
Participants | 156 | 114
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Multiple imputation was used to estimate missing data for the 9-month assessment. Ten datasets were imputed using Multivariate Imputation by Chained Equations. Using SAS v9.1 PROC MI, the complete datasets were analyzed using complete data methodology-in this case, logistic regression-and the results pooled; Test type: Non-Inferiority or Equivalence — Power analysis shows that sample size provided power of at least .80 to detect estimated differences; p = .002, t-test, 1 sided — [p-value comment as in outcome 1, analysis 1]; t(181) = 2.9

3. Secondary Outcome: Number of Participants in the Action or Maintenance Stage for Using Effective Methods to Prevent Depression.
Description: Depression prevention was defined as: "Using effective methods to keep depression from occurring, or if it does occur, to keep it as mild and brief as possible." Effective methods were: 1) controlling negative thinking; 2) engaging in healthy, pleasant activities; 3) practicing stress management; 4) exercising; and 5) getting professional help when needed. Patients who reported that they were not currently practicing depression prevention and had no intention of doing so in the next 6 months were classified in the precontemplation stage; those who intended to practice depression prevention in the next 6 months or next 30 days were classified in the contemplation or preparation stage, respectively; those who had been practicing depression prevention for less than 6 months were in the action stage, and those who had been practicing for more than 6 months were in maintenance. This outcome represents the number of participants in the action or maintenance stage at 9 months follow-up.
Time Frame: 9 months
Population: Multiple imputation
Measure: Number; unit: Participants
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 443 | 459
Participants | 339 | 324
Statistical Analysis 1: Comparison: Intervention vs Usual Care; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — Power analysis shows that sample size provided power of at least .80 to detect estimated differences; p = .04, t-test, 1 sided — [p-value comment as in outcome 1, analysis 1]; t(153) = 1.8

4. Secondary Outcome: Number Participants Without Major Depression at Baseline Who Experienced the Onset of Major Depression During Follow-up
Description: At baseline and follow-up, Major Depression was assessed using 9-item depression module of the Primary Care Evaluation of Mental Disorders Patient Health Questionnaire-PHQ-9 (Spitzer, Kroenke, & Williams, 1999). In this analysis, Major Depression was assessed among participants not meeting criteria for major depression at baseline.
Time Frame: 9 months
Population: Multiple imputation
Measure: Number; unit: Participants
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 369 | 385
Participants | 49 | 72
Statistical Analysis 1: Comparison: Intervention vs Usual Care; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — Power analysis shows that sample size provided power of at least .80 to detect estimated differences; p = .07, t-test, 1 sided — [p-value comment as in outcome 1, analysis 1]; t(57) = 1.5

5. Secondary Outcome: Number of Participants Taking Prescribed Antidepressant Medication (Medication Adherence)
Description: At 9 months follow-up, participants who had been prescribed antidepressant medication were asked if they had started and were still taking it. Participants who were taking their medication or had stopped with their doctor's advice were considered to be adherent.
Time Frame: 9 months
Population: Multiple imputation
Measure: Number; unit: Participants
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 195 | 194
Participants | 121 | 100
Statistical Analysis 1: Comparison: Intervention vs Usual Care; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — Power analysis shows that sample size provided power of at least .80 to detect estimated differences; p = .05, t-test, 1 sided; t(94) = 1.5

6. Secondary Outcome: Change in Physical Functioning
Description: Physical functioning was assessed using the Physical Functioning, Role Functioning, Health Perceptions, and Pain subscales of the 20-item Medical Outcomes Study Short Form survey (SF-20) (Stewart, Hays, & Ware, Jr., 1988). (SF-20 subscales assessing mental health and social functioning were omitted to get a purer measure of physical functioning). Physical functioning was computed by taking the mean of the four subscales after each was linearly transformed to range from 0-100. The change scores reported here are the difference between the physical functioning scores at baseline and 9 months (i.e., 9 months minus baseline). Change scores range from -100 to +100, with higher positive scores indicating more improvement in physical functioning.
Time Frame: Baseline, 9 months
Population: Multiple imputation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 443 | 459
units on a scale | 3.1 (16.5) | 1.6 (16.3)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Power analysis shows that sample size provided power of at least .80 to detect estimated differences; p = .13, t-test, 1 sided — [p-value comment as in outcome 1, analysis 1]; t(123) = 1.2

ADVERSE EVENTS:
Time Frame: 36 months
Arm/Group | Intervention | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/443 | 0/459
Other Adverse Events (participants affected / at risk) | 0/443 | 0/459

LIMITATIONS AND CAVEATS:
1. There was only a single follow up assessment administered at 9 months post-baseline.
2. The study attrition rate was > 30%.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No